CLINICAL TRIAL: NCT01249586
Title: E-learning as a Complement to Traditional Teaching of Blindness Prevention
Brief Title: E-learning: Teaching of Blindness Prevention
Acronym: ELBPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinica Oftamologica Zona Sul (Other)
Other Study IDs: ELBPS
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Teaching Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Traditional teaching (Placebo Comparator): A traditional class of blindness prevention.
  Interventions: Other: E-learning

INTERVENTIONS:
Other: E-learning — A traditional class of blindness prevention plus an additional e-learning material. The e-learning material included a PDF article about blindness prevention. This material was e-mailed one week before the traditional class.

SUMMARY:
E-learning material increases the student knowledge level before the traditional class of blindness prevention and help to fix this information a short period (one month) after the class.

ELIGIBILITY:
Inclusion Criteria:

* being a medical student matriculated in the course of ophthalmology. This course is taught to fourth-year students at State University of Campinas.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Immediate pretest score

SECONDARY OUTCOMES:
One-month posttest score
Immediate posttest score.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinics Hospital of the State University of Campinas, Campinas, São Paulo, Brazil